CLINICAL TRIAL: NCT00747695
Title: A Pharmacokinetic and Safety Study of Single and Multiple Doses of Rabreprazole in Pediatric Patients With GERD 1 to 11 Years Old, Inclusive
Brief Title: A Pharmacokinetic and Safety Study of Single and Multiple Doses of Rabreprazole in Pediatric Patients With Gastroesophageal Reflux Disease (GERD) 1 to 11 Years Old, Inclusive
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Eisai Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013945
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2011-01

CONDITIONS: GERD
Keywords: Pediatric Pharmacokinetics; Pediatric Pharmacodynamics; Rabeprazole; Pediatric GERD; Aciphex
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole

INTERVENTIONS:
Drug: Rabeprazole sodium

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics, pharmacodynamics and safety of rabeprazole after single and multiple daily administration in children between the ages of 1 and 11 years, inclusive, with GERD.

DETAILED DESCRIPTION:
This is an open-label (both the physician and the patient know the name of the study medication), multi-center, Phase 1 study, consisting of 2 parts. The first part of the study will be non-randomized, all patients will receive the same dose. In the second part of the study, patients will be randomized (study medication assigned by chance) into 2 dose groups. The purpose of the study is to evaluate the pharmacokinetics, pharmacodynamics (clinical global impressions and formulation palatability) and safety of rabrepazole after single and multiple daily administration at 2 dose levels in children between the ages of 1 and 11 years, inclusive, with GERD. As this study is an exploratory assessment of the pharmacokinetics, pharmacodynamics and safety of rabeprazole in children, no formal hypothesis testing is applied. Safety and tolerability, including monitoring of adverse events, clinical laboratory results, physical examination, vital signs and ECG measurements, will be evaluated throughout the study. Patients will receive rabeprazole sodium as single daily oral doses for 5 successive days as a bead formulation. Patients in the first part of the study will receive single and multiple daily every 24 hours doses of 0.14 mg/kg, using increments of 1 mg dose. Safety and pk data from part 1 of the study will determine the 2 dosages to be studied in part 2 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Boy and girls and a minimum weight of 10 kg with endoscopically proven GERD including an endoscopic examination as part of their diagnostic evaluation
* Patients who have been treated with, or are currently receiving a proton pump inhibitor (PPI), H2 blockers, or antacids are eligible (as long as they can go off antacids for 24 hours, and PPIs and H2 blockers for 3 days prior to dosing, except for cimetidine, which must be discontinued for at least 7 days prior to dosing) and remain off these medications for the treatment period
* Patients who are generally healthy, other than the presence of GERD, with the exception of the following: Patients with stable asthma/reactive airway disease or cystic fibrosis-dependent GERD symptoms on stable treatment regimens or subjects on stable doses of allergy and attention deficit disorder medicines.

Exclusion Criteria:

* Patients who have a history of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders, lipid abnormalities, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the subject or that could interfere with the interpretation of the study results
* Primary pulmonary or ENT symptoms
* Presence of "warning signals", suggesting cause of vomiting/regurgitation other than GERD
* History of primary esophageal motility disorders or systemic condition affecting the esophagus
* History of eosinophilic esophagitis, persistent milk protein allergy, or allergic gastroenteropathy
* History of or current presence of peptic ulcers
* Current presence of Helicobacter pylori
* History of definitive acid-lowering surgery
* Significant arrhythmias.

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2008-03; Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic, pharmacodynamic and safety parameters of rabeprazole will be listed and summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.